CLINICAL TRIAL: NCT06024928
Title: Short Use of Automated Insulin Delivery (AID) for Basal Insulin Titration in Type 2 Diabetes: A Pilot Study
Brief Title: Automated Insulin Delivery (AID) for Basal Insulin Titration in Type 2 Diabetes
Acronym: AID-BIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anas El Fathi, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 230316; 1R01DK133148 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes
Keywords: Automated Insulin Delivery (AID); Continuous Glucose Monitor (CGM); Tandem t:slim Insulin Pump with Control-IQ Technology (CIQ); Basal Insulin Titration (BIT)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled parallel design trial where participants will be randomized 1:1 to either a control group or an experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Automated Insulin Delivery in the Basal Insulin Titration Phase (Experimental): Participants will use Automated Insulin Delivery (AID) for 10 days in the Basal Insulin Titration (BIT) Phase. This group will then return to their original home therapy (basal insulin using pen) using the new setting in the Maintenance Phase (MP) with a blinded CGM. The total daily insulin (TDI) requirement during the BIT Phase will be translated to a basal insulin dose.
  Interventions: Device: Control-IQ use in Type 2 Diabetes under basal insulin injections
- Standard Care with Study Continuous Glucose Monitor (No Intervention): Participants will use a study Continuous Glucose Monitor (CGM) along with their original home therapy and will be contacted by a study physician as per standard care to adjust their insulin doses if needed. This group will then transition into a 10-day Maintenance Phase (MP) using a blinded CGM, where the basal dose will be maintained.

INTERVENTIONS:
Device: Control-IQ use in Type 2 Diabetes under basal insulin injections — Testing the safety and feasibility of using Automated Insulin Delivery (AID) in people with Type 2 Diabetes under basal insulin injections to achieve safe and fast basal insulin titration.
  Other Names: Tandem Diabetes Care
  Arms: Automated Insulin Delivery in the Basal Insulin Titration Phase

SUMMARY:
The purpose of this clinical trial is to test the safety and feasibility of using an Automated Insulin Device (AID) in people with Type 2 Diabetes under basal insulin injections to achieve safe and fast basal insulin titration. Participants will be randomized to either the control group or the experimental group. If in the experimental group, the participant will use an insulin pump with Control-IQ Technology (Tandem Diabetes Care) for ten days. Researchers will compare the glycemic control of the experimental group to the control group.

DETAILED DESCRIPTION:
The study will involve 20 people with Type 2 Diabetes who are 18 years or older. The study will be performed at the University of Virginia (UVA), with screening procedures taking place either virtually or at the Clinical Research Unit (CRU) at UVA. All participants will undergo a 10-day run-in phase with a blinded Dexcom Generation 6 Continuous Glucose Monitor (CGM). Participants will be randomized (1:1) to either the Control (CTR) Group or the Experimental (EXP) Group. In the EXP Group, participants will use an Automated Insulin Device (AID) for 10 days in the Basal Insulin Titration (BIT) Phase then return to their original therapy (basal insulin using pen) using the new setting in the Maintenance Phase (MP). The total daily insulin (TDI) requirement during the BIT Phase will be translated to a basal insulin dose. During the same 10 days, in the CTR group, participants will use an unblinded CGM and will be contacted by a study physician as per standard care to adjust their insulin doses if needed. Both groups will then go into a 10-days maintenance period using a blinded CGM. Outcomes will be measured in the last 7 days of the BIT and Maintenance Phases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 years old at time of consent.
2. Clinical diagnosis, based on investigator assessment, of type 2 diabetes for at least one year.
3. HbA1c ≥ 7.5%.
4. Currently using an approved long-acting insulin for at least two months (e.g., insulin glargine, insulin degludec)
5. If using a CGM, willingness to wear an additional study CGM during the duration of the study.
6. Access to the internet and willingness to upload data during the study as needed.
7. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females who self-report that they are of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
8. Willingness to remain on same dose of non-insulin glucose-lowering agent during the trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, sulfonylureas and naturaceuticals).

Exclusion Criteria:

1. Currently using an approved intermediate (e.g., insulin NPH) or rapid insulin for at least six months (e.g., insulin aspart, insulin lispro, insulin regular).
2. Currently being treated for a seizure disorder.
3. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol, such as but not limited to, the following examples:

   1. Inpatient psychiatric treatment in the past 6 months
   2. Presence of a known adrenal disorder
   3. Uncontrolled thyroid disease
4. Currently pregnant or intent to become pregnant during the trial.
5. Currently breastfeeding.
6. Anticipated surgical, interventional procedures or prolonged periods of fasting during this study.
7. History of hypoglycemia unawareness.
8. On a non-stable dose of non-insulin glucose-lowering agent prior to the trial (including metformin/biguanides, GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, sulfonylureas and naturaceuticals) as defined by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
System Testing survey | 14 days
  Receiving feedback from the participants regarding system functionality.
Percent Time in Range | 14 days
  The percent of time spent within glycemic range of 70 to 180 mg/mL.

SECONDARY OUTCOMES:
Percent Time Below Range | 14 days
  The percent of time spent below 70 mg/mL.
Percent Time Above Range | 14 days
  The percent of time spent above 180 mg/mL.
Percent Time in Tighter Range | 14 days
  The percent of time spent within glycemic range of 70 to 140 mg/mL.
Percent Time Below Range (Hypoglycemia) | 14 days
  The percent of time spent below 54 mg/mL.
Percent Time Above Range (Hyperglycemia) | 14 days
  The percent of time spent above 250 mg/mL.
Mean glucose reading measured by Continuous Glucose Monitor (CGM) | 14 days
  Glucose variability measured by coefficient of variation.

CONTACTS AND LOCATIONS:
Overall Officials: Anas El Fathi, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (2):
- United States (2):
  - VA Maryland Health Care System, Baltimore, Maryland
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available after the primary publications of the study.
Access Criteria: The Data Sharing Agreements will be formulated by the study team.